CLINICAL TRIAL: NCT01412411
Title: Appropriate Complementary Feeding Strategies in Infants: An Evaluation of Various Strategies to Assess the Growth and Health of the Infants.
Brief Title: Appropriate Complmentary Feeding Strategies in Infants
Acronym: CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); European Union (Other)
Responsible Party: Dr Aziz Abdul Rehman Jiwani, The Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 480/Peds-ERC-05
Record Dates: First submitted 2011-08-03; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2008-03

CONDITIONS: Anemia
Keywords: Anemia; Growth; Infants; Focus of the study is to assess the level of anemia and growth indicators among the infants
MeSH Terms: conditions — Anemia | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nutrition Education plus Multiple Micronutrient Fortification (Active Comparator): In this group along with the nutritional education, multiple micronutrient fortification was given in the form of Sprinkles
  Interventions: Dietary Supplement: Multiple micronutrient fortification plus Nutrition Education
- OIS plus Nutritional Eductaion (Active Comparator): In this group, along with the nutritional education, Oral Iron Supplementation was given.
  Interventions: Dietary Supplement: Oral Iron Supplementation along with Nturition Eductaion
- Nutrition Education Group (Active Comparator): This is group was followed for the growth of the child and was given Nutritional Education to children's mothers.
  Interventions: Behavioral: Nutritionl Education

INTERVENTIONS:
Behavioral: Nutritionl Education — to assess the change in behaviour
  Arms: Nutrition Education Group
Dietary Supplement: Oral Iron Supplementation along with Nturition Eductaion
  Arms: OIS plus Nutritional Eductaion
Dietary Supplement: Multiple micronutrient fortification plus Nutrition Education
  Arms: Nutrition Education plus Multiple Micronutrient Fortification

SUMMARY:
The purpose of this study has been to understand the prevalence of under nutrition and develop effective interventions for improving growth and micronutrient status of infants receiving complementary foods.

In this community based randomized clinical trial, the nutrition education package implemented aimed to improve hematological parameters including the micronutrient status and to see effect on growth indicators.

DETAILED DESCRIPTION:
Transition from exclusive breast feeding to complementary feeding poses many challenges as the demand for nutrients necessary for optimum growth and development increases steadily. Malnutrition and micronutrient malnutrition can be inter-generational and affect pregnant mothers and consequently the baby may be born with deficient micronutrient stores, especially those of iron. This deficiency can be further exacerbated by sub-optimal practices of breast feeding. Globally, iron deficiency is the most common cause of anemia estimated to affect nearly 2 billion people especially preschool children. In Pakistan, 56 % of children under the age of five years are estimated to have iron deficiency anemia and 13 % are also severely malnourished. These deficiencies affect not only physical growth but also mental development with significant impact on immunity and increased burden of infections. It is uncertain what the most appropriate intervention strategy is and a wide range of options are mentioned including dietary diversification through nutrition education, provision of fortified foods, iron supplementation and home-based fortification of complementary foods with micronutrient powders such as Sprinkles.

In an effort to understand the prevalence of under nutrition and develop effective interventions for improving growth and micronutrient status of infants receiving complementary foods, I undertook a prospective community-based randomized controlled efficacy trial in a representative urban population of Karachi. Infants and mothers were identified after birth and enrolled in the study to receive one of the interventions through community health workers at the age of six months. The enrolled infants were placed in three groups - defined as Nutr Education (Nutr Edu), Oral iron supplementation (OIS) and Multiple micronutrient fortification (MMF). Nutrition education component was common to all the groups. Through nutritional education sessions held in the community, dietary diversification along with continuation of breast feeding was stressed to enhance the intake of diet, rich in iron, and other micronutrients. A cohort of 451 infants (177 in group Nutr Edu, 141 in group OIS and 133 in MMF) were followed for three months (till the end of treatments) for growth, micronutrient status, and morbidity rate and thereafter followed for another three months to evaluate anthropometric parameters.

ELIGIBILITY:
Inclusion Criteria:

* All children between the age of 6 months to 8 months.

Exclusion Criteria:

* Children who are sick to an extent that cannot take anythign oral were excluded from this study.

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Anemia | 12 months
  To assess the impact of supplementation and multiple micronutrient fortification in comparison to nutritional education strategy to assess the biochecmical and growth indicators

SECONDARY OUTCOMES:
Compliance to intake of study medicines | 12 months
  Compliance was checked to ensure that subjects are taking study medicines properly.
Morbidity Assessment | 12 months
  Subjects were assessed on fortnighty basis to see any change in the morbidity.
Developmental Assessment | 12 months
  Subjects were assessed on monthly developmental milestones among the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz AJ Abdul Rehman Jiwani, MBBS, PhD, Principal Investigator — Aga Khan University; Zulfiqar ZB Bhuta, MBBS, MCPS (Peds), FCPS (Peds), Study Chair — Aga Khan University
Locations (1):
- Bilal Colony Centre, Karachi, Sindh, Pakistan